CLINICAL TRIAL: NCT01496066
Title: A Prospective Randomized Controlled Multi-Center Clinical Study to Evaluate the Safety and Effectiveness of the Light Adjustable Lens (LAL) in Subjects With Pre-Existing Corneal Astigmatism
Brief Title: Calhoun Vision Light Adjustable Lens (LAL) in Subjects With Pre-Existing Corneal Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Calhoun Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSP-002-03
Record Dates: First submitted 2011-12-15; First posted 2011-12-21 (Estimated); Results first posted 2018-03-05 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-05

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: Phase 3 medical device study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LAL (Experimental): LAL implanted
  Interventions: Device: LAL (Light Adjustable Lens) and Light Deliver Device (LDD)
- Monofocal control (Active Comparator): Monofocal control IOL implanted
  Interventions: Device: Monofocal control IOL

INTERVENTIONS:
Device: LAL (Light Adjustable Lens) and Light Deliver Device (LDD) — LAL implanted and adjusted with LDD
  Arms: LAL
Device: Monofocal control IOL — Commercially available monofocal intraocular lens (IOL)
  Arms: Monofocal control

SUMMARY:
The purpose is to evaluate the Calhoun Vision Light Adjustable Lens (LAL) and Light Delivery Device (LDD) for reducing astigmatism and improving uncorrected vision after implantation.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing cataract surgery and be willing to have LAL or commercially available IOL implanted
* Pre-operative regular corneal astigmatism of >= 0.75 diopters and <= 2.0 diopters
* Best spectacle corrected visual acuity reduced to 20/40 or worse with or without glare
* Projected best spectacle corrected visual acuity of 20/20 or better
* Clear intraocular media other than cataract
* Potentially good vision in fellow eye
* Fully dilated pupil of >= 7.0 mm

Exclusion Criteria:

* Zonular laxity or dehiscence
* Pseudoexfoliation
* Age related macular degeneration
* Retinal degenerative disorder
* Diabetes with any evidence of retinopathy
* Glaucomatous optic neuropathy, uveitis, significant anterior segment pathology, keratoconus
* Corneal dystrophy, previous corneal or intraocular surgery
* Complications during cataract surgery
* Serious co-morbid conditions
* Systemic medications that my increase UV sensitivity
* Irregular astigmatism

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2011-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Vold Vision, Fayetteville, Arkansas
  - Jules Stein Eye Institute, Los Angeles, California
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - Newsom Eye, Sebring, Florida
  - Arbor Centers for Eye Care, Orland Park, Illinois
  - Eye Surgeons of Indiana, Indianapolis, Indiana
  - Jones Eye Clinic, Sioux City, Iowa
  - Discover Vision & Laser Center, Leawood, Kansas
  - Minnesota Eye Consultants, PA, Bloomington, Minnesota
  - Ophthalmology Consultants, Ltd., St Louis, Missouri
  - EyeSight Ophthalmic Services, PA, Somersworth, New Hampshire
  - Carolina Vision Center, Fayetteville, North Carolina
  - Cleveland Eye Clinic, Brecksville, Ohio
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Eye Consultants of Texas, Grapevine, Texas
  - Focal Point Vision, San Antonio, Texas
  - Hoopes Vision, Draper, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- LAL Implant: LAL implanted
  LAL (Light Adjustable Lens) and Light Deliver Device (LDD): LAL implanted and adjusted with LDD
Period: Overall Study
Arm/Group | LAL Implant | Monofocal Control
Started | 403 | 197
Completed | 391 | 188
Not Completed | 12 | 9
Not completed — Lost to Follow-up | 8 | 5
Not completed — Explant | 3 | 0
Not completed — Death | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LAL Implant | Monofocal Control | Total
Number analyzed (Participants) | 403 | 197 | 600
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (7.9) | 66.6 (7.2) | 66.2 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 242 | 102 | 344
  Male | 161 | 95 | 256
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 7 | 25
  Not Hispanic or Latino | 385 | 190 | 575
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 15 | 6 | 21
  White | 383 | 188 | 571
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Right Eye [Number; unit: Eyes] | 226 | 96 | 322
Left Eye [Number; unit: Eyes] | 177 | 101 | 278

OUTCOME MEASURES:

1. Primary Outcome: Percent Reduction in Manifest Cylinder
Description: Percent reduction in manifest cylinder from Pre-Adjustment (LAL) or 17-21 days post-op (control) to 6 months postop. Manifest cylinder refers to only the astigmatic or cylindrical component of an ophthalmic manifest refraction. For example if someone had a refraction of +0.50-1.00x090, the -1.00 is the manifest cylinder component. The reduction of the manifest cylinder is determined from Pre-Adjustment (LAL) or 17-21 days post-op (control) to 6 months postop.
Time Frame: 6 months
Population: ITT. Only eyes that had cylinder in the range of treatment (>=0.75 D) were included in the analysis. Therefore the number of participants analyzed for this outcome measure will not match the overall number of participants in the study.
Measure: Mean (95% Confidence Interval); unit: percent reduction in manifest cylinder
Groups:
- Light Adjustable Lens Implanted: Randomized to have the Light Adjustable Lens implanted
- Control IOL Implanted: Randomized to have the monofocal control IOL implanted
Arm/Group | Light Adjustable Lens Implanted | Control IOL Implanted
Number analyzed (Participants) | 286 | 126
percent reduction in manifest cylinder | 74.6 [71.1 to 78.1] | 19.9 [10.9 to 28.9]

2. Primary Outcome: Percent Absolute Reduction in MRSE
Description: Percent absolute reduction in Manifest Refraction Spherical Equivalent (MRSE) from Pre-Adjustment (LAL) or 17-21 days post-op (control) to 6 months postop. It is used to describe an ophthalmic refraction with one number. It is defined as the (sphere)+ 0.5(cylinder). So, if you had a refraction of +1.00-1.00x090 the MRSE would be +0.50, the +1.00 is the sphere and the -1.00 is the cylinder in this example. If you had a refraction of +0.25-1.50x145 the MRSE would be -0.50. The absolute value of the MRSE is taken and its reduction is calculated from Pre-Adjustment (LAL) or 17-21 days post-op (control) to 6 months postop.
Time Frame: 6 months
Population: ITT. Any eyes that had an MRSE of zero at Pre-Adjustment were excluded since it is not possible to divide by zero. Therefore the number participants analyzed for this outcome will differ from the number of overall participants in the study.
Measure: Mean (95% Confidence Interval); unit: percentage of reduction in MRSE
Groups:
- Light Adjustable Lens: Eyes randomized to have Light Adjustable Lens implanted
- Monofocal Control IOL: Eyes randomized to have monofocal control IOL implanted
Arm/Group | Light Adjustable Lens | Monofocal Control IOL
Number analyzed (Participants) | 380 | 166
percentage of reduction in MRSE | 51.5 [43.8 to 59.1] | 10.4 [-3.8 to 24.7]

3. Primary Outcome: Rotation of LAL Landmark Meridian to Anatomical Landmark at Pre-Adjustment and 6 Months Postop
Description: Number (%) of eyes with rotation of LAL meridian of ≤ 5 degrees from Pre-Adjustment to 6 months postop. This endpoint was achieved by taking dilated anterior segment photographs of the LAL at Pre-Adjustment and 6 months postop. The angular difference between a landmark on the LAL and an anatomical landmark on the subjects eye was measured. The same landmarks on the LAL and the subjects eye were used at each time point. The angular difference between the two time points was then determined.
Time Frame: 6 months
Population: ITT: The overall number of participants analyzed differs from the other outcome measures because some photographs were unusable due to inadequate lighting, user error, or equipment failure.
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Groups:
- Light Adjustable Lens: Eyes randomized to be implanted with the Light Adjustable Lens
Arm/Group | Light Adjustable Lens
Number analyzed (Participants) | 358
percentage of eyes | 96.1 [93.5 to 97.8]

4. Secondary Outcome: Uncorrected Visual Acuity 20/20 or Better
Description: Percent of eyes with UCVA of 20/20 or better in the LAL treatment group at 6 months postoperatively was calculated to determine if it is significantly greater than the percent of eyes with UCVA of 20/20 or better in the monofocal control group at 6 months postoperatively.
Time Frame: 6 months
Population: ITT
Measure: Number; unit: percentage of eyes
Groups:
- Light Adjustable Lens: Randomized to have the Light Adjustable Lens implanted
- Monofocal Control IOL: Randomized to have a Monofocal control IOL implanted
Arm/Group | Light Adjustable Lens | Monofocal Control IOL
Number analyzed (Participants) | 391 | 193
percentage of eyes | 70.1 | 36.3
Statistical Analysis 1: Comparison: Light Adjustable Lens vs Monofocal Control IOL; Test type: Superiority; p < .0001, Chi-squared

5. Secondary Outcome: Mean Reduction in Cylinder by Cylinder Adjustment Stratum (0.75D-1.25D)
Description: Percent reduction in absolute manifest cylinder in the LAL treatment group was calculated to determine if it is significantly greater than the percent reduction in absolute cylinder in the monofocal control group at 6 months postoperatively compared to pre-adjustment in the LAL group/17-21 days postoperative in the control group. Results were to be evaluated for each cylinder adjustment stratum (0.75-1.25 D and 1.50-2.00 D) separately.
Time Frame: 6 months
Population: Participants with eyes in ITT with 0.75-1.25 D cylinder prior to light treatment
Measure: Mean (Standard Deviation); unit: percent reduction in cylinder
Groups:
- Monofocal Control IOL: Randomized to have the monofocal control IOL implanted
Arm/Group | Light Adjustable Lens | Monofocal Control IOL
Number analyzed (Participants) | 203 | 90
percent reduction in cylinder | 73.4 (33.1) | 18.6 (57.0)
Statistical Analysis 1: Comparison: Light Adjustable Lens vs Monofocal Control IOL; Test type: Superiority; p < .0001, t-test, 2 sided

6. Secondary Outcome: Mean Reduction in Cylinder by Cylinder Adjustment Stratum (>1.25D)
Description: Percent reduction in absolute manifest cylinder in the LAL treatment group was calculated to determine if it is significantly greater than the percent reduction in absolute cylinder in the monofocal control group at 6 months postoperatively compared to Pre-Adjustment in the LAL group/17-21 days postoperative in the control group.
Time Frame: 6 months
Population: Participants with eyes in ITT with >1.25 D of cylinder prior to light treatment
Measure: Mean (Standard Deviation); unit: percent reduction in cylinder
Arm/Group | Light Adjustable Lens | Monofocal Control IOL
Number analyzed (Participants) | 83 | 36
percent reduction in cylinder | 77.5 (20.7) | 23.1 (32.3)
Statistical Analysis 1: Comparison: Light Adjustable Lens vs Monofocal Control IOL; Test type: Superiority; p < .0001, t-test, 2 sided

7. Secondary Outcome: Percent Absolute Reduction in Manifest Refraction Spherical Equivalent (MRSE) for Eyes With <0.75 D Cylinder Postoperatively
Description: For eyes with <0.75 D of cylinder at pre-adjustment (LAL)/17-21 days (control group), percent mean absolute reduction in MRSE by subject in the LAL treatment group was calculated to determine if it is significantly greater than the percent reduction in mean absolute MRSE in the monofocal control group at 6 months postoperatively compared to pre-adjustment in the LAL group/17-21 days postoperative in the control group.
Time Frame: 6 months
Population: Participants with eyes in ITT with <0.75 D of cylinder prior to light treatment
Measure: Mean (Standard Deviation); unit: percent absolute reduction in MRSE
Arm/Group | Light Adjustable Lens | Monofocal Control IOL
Number analyzed (Participants) | 100 | 53
percent absolute reduction in MRSE | 55.2 (76.3) | 27.2 (75.2)
Statistical Analysis 1: Comparison: Light Adjustable Lens vs Monofocal Control IOL; Test type: Superiority; p = .0318, t-test, 2 sided

8. Secondary Outcome: Mean BSCVA
Description: Mean BSCVA for the "best case" cohort (no macular problems) at 6 months postoperatively was compared between the LAL treatment group and the monofocal control group. Endpoint success was to be achieved if the difference in mean BSCVA between the LAL cohort and the monofocal control group is within 1 line (0.1 LogMAR) (non-inferiority margin or delta).
Time Frame: 6 months
Population: ITT population best case cohort with no macular problems
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Light Adjustable Lens | Monofocal Control IOL
Number analyzed (Participants) | 390 | 191
LogMAR | -0.066 (0.083) | -0.029 (0.090)
Statistical Analysis 1: Comparison: Light Adjustable Lens vs Monofocal Control IOL; Test type: Equivalence — a two-group t-test of equivalence in means was used; Mean Difference (Final Values) = -0.04, 99% CI 2-sided [-0.06 to -0.02]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Light Adjustable Lens | Monofocal Control IOL
All-Cause Mortality (participants affected / at risk) | 1/403 | 4/197
Serious Adverse Events (participants affected / at risk) | 42/403 | 10/197
Other Adverse Events (participants affected / at risk) | 292/403 | 125/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Light Adjustable Lens (N=403) | Monofocal Control IOL (N=197)
Herpetic Keratouveitis (Eye disorders) | 1 (1) | 0 (0)
Persistent Induced Tritan Color Anomaly (Eye disorders) | 2 (2) | 0 (0)
Cystoid Macular Edema (Eye disorders) | 3 (3) | 3 (3)
Endophthalmitis (Eye disorders) | 1 (1) | 0 (0)
Horseshoe retinal tear with vitreous hemorrhage (Eye disorders) | 1 (1) | 1 (1)
Hypopyon (Eye disorders) | 1 (1) | 0 (0)
Surgical complication (Eye disorders) | 1 (1) | 0 (0) — Surgical complication including anterior segment bleeding, vitreous loss, and posterior capsule and zonular rupture
Anxiety (Nervous system disorders) | 1 (1) | 0 (0)
Blood clots due to lymphoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Broken blood vessel in brain (Vascular disorders) | 0 (0) | 1 (1)
Broken wrist (General disorders) | 1 (1) | 0 (0)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chest pain with pacemaker (Cardiac disorders) | 1 (1) | 0 (0)
Heart palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Heart surgery (Cardiac disorders) | 1 (1) | 0 (0)
Hospitalization due to cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Hospitalization due to concussion with subdural hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hospitalization due to emphysema/COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hospitalization due to infection after knee surgery (Infections and infestations) | 1 (1) | 0 (0)
Hospitalization due to syncope (General disorders) | 1 (1) | 0 (0)
Hospitalization for colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hospitalization due to low blood pressure and syncope (General disorders) | 1 (1) | 0 (0)
Hospitalization due to dizziness (General disorders) | 1 (1) | 0 (0)
Kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Liver cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neuroendocrine tumors (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Stroke (Vascular disorders) | 2 (2) | 0 (0)
Transient ischemic attack (Vascular disorders) | 0 (0) | 1 (1)
Triple bypass surgery (Cardiac disorders) | 0 (0) | 1 (1)
Secondary surgical intervention (Eye disorders) | 7 (7) | 1 (1)
Phytotoxic retinal damage causing temporary loss of BSCVA (Eye disorders) | 1 (1) | 0 (0)
Persistent induced erythropsia (Eye disorders) | 1 (1) | 0 (0)
Persistent unanticipated increase refractive error (Eye disorders) | 5 (5) | 0 (0)
Intraoperative capsular tear (Eye disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Light Adjustable Lens (N=403) | Monofocal Control IOL (N=197)
Anterior chamber cells (Eye disorders) | 43 (43) | 21 (21)
Anterior chamber flare (Eye disorders) | 19 (19) | 11 (11)
Blurred vision (Eye disorders) | 31 (31) | 19 (19)
Corneal edema central (Eye disorders) | 25 (25) | 13 (13)
corneal edema wound (Eye disorders) | 43 (43) | 14 (14)
Posterior capsular opacity (Eye disorders) | 51 (51) | 26 (26)
Raised IOP not requiring treatment (Eye disorders) | 32 (32) | 2 (2)
Raised IOP requiring treatment (Eye disorders) | 26 (26) | 14 (14)
Superficial punctate keratitis (Eye disorders) | 22 (22) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No